CLINICAL TRIAL: NCT04729569
Title: Gingival Response and Marginal Adaptation of Zirconia Crowns With Two Subgingival Margin Designs: A Randomized Clinical Trial
Brief Title: Gingival Response and Marginal Adaptation of Zirconia Crowns With Two Subgingival Margin Designs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Hassan El-Khayat, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 161020
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Gingival Recession, Localized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tested finish line preparation (Other): Feather edge finish line preparation (Intervention)
  Interventions: Procedure: Feather edge finish line preparation
- Comparator finish line preparation (Active Comparator): Deep chamfer finish line preparation (Comparator)
  Interventions: Procedure: Deep chamfer finish line preparation

INTERVENTIONS:
Procedure: Feather edge finish line preparation — Tooth preparation with feather edge finish line will be done to posterior teeth to receive all ceramic full coverage zirconia crowns.
  Arms: Tested finish line preparation
Procedure: Deep chamfer finish line preparation — Tooth preparation with deep chamfer finish line will be done to posterior teeth to receive all ceramic full coverage zirconia crowns.
  Arms: Comparator finish line preparation

SUMMARY:
The aim of the study is to evaluate the effect of feather edge finish line and deep chamfer finish line on gingival position, bleeding on probing and marginal adaptation.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effect of feather edge finish line and deep chamfer finish line on gingival position, bleeding on probing and marginal adaptation.

Gingival bleeding on probing will be evaluated before treatment. Preparation for all ceramic full coverage restoration will be performed according to manufacturer instructions by one operator. Type of finish line (whether feather edge or deep chamfer finish line) will be selected randomly according to a computer generated randomization list. Restorative margins will be placed subgingivally. Zirconia crowns will be fabricated for the prepared teeth and cemented using resin luting agent. At 6 months and 12 months after the cementation, restorative margin position relative to the gingival margin will be recorded. Bleeding on probing and marginal adaptation will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years to 50 years old
* Dentate patients planned for a single full coverage restoration in the posterior area.
* Patients with no active periodontal disease.
* >2mm of keratinized tissue

Exclusion Criteria:

* Smoking (>10 cigarettes a day)
* Substance abuse history
* Patients with poor oral hygiene and high caries index
* Patients suffering from abnormal occlusal habits for example clenching or bruxism
* Local or systemic disease (endocrine, renal, hematologic, hepatic, immunosuppressive)
* Current steroid/chemotherapy
* Head and neck irradiation
* Pregnancy
* Inability or unwillingness to return for follow up visits.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Position of the margin of the restoration in relation to the gingival margin position | 1 year
  Scoring proposed by Paniz et al classified into either subgingival (not visible), equigingival (slightly visible) and supragingival (visible)

SECONDARY OUTCOMES:
Bleeding on probing | 1 year
  Scoring following Ainamo and Bay gingival bleeding index

OTHER OUTCOMES:
Marginal adaptation | 1 year
  Evaluation using Modified USPHS criteria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] El-Khayat H, Anwar EM, Nabil O, Aboushahba M. Gingival Recession and Marginal Adaptation of Zirconia Crowns with Two Subgingival Margin Designs: A Randomized Clinical Trial. J Contemp Dent Pract. 2025 Aug 1;26(8):767-775. doi: 10.5005/jp-journals-10024-3932. PMID 41145363